CLINICAL TRIAL: NCT06784635
Title: The Effect of Remote Treatment on Medical Provider Creative Thinking and Patient Disclosure
Acronym: MED-CREATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayoub Bouguettaya (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor-Investigator, Ayoub Bouguettaya, Principal Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00003845
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Focus is on Behavior of Health Professionals Generally
Keywords: Patient disclosure; human-computer interaction; social psychology; health psychology; healthcare delivery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online interaction (Experimental): Participant allocated to this arm will meet online, although they will be in the same building. They will have a conversation over an encrypted video platform.
  Interventions: Behavioral: Online interaction
- In person interaction (Experimental): Participant allocated to this arm will meet in person, in the same room. They will have a conversation face to face in an office setting.
  Interventions: Behavioral: In person

INTERVENTIONS:
Behavioral: In person — Participant dyads will meet in person for a mock clinical interview, seated at a desk opposite their counterpart. They will be in an office setting. There will be a sham white noise and lamp device placed on the desk.
  Arms: In person interaction
Behavioral: Online interaction — Participant dyads will meet online in a mock clinical interview, via an encrypted video call, seated at a desk. They will be in an office setting. There will be a sham white noise and lamp device placed on the desk.
  Arms: Online interaction

SUMMARY:
The investigators will be doing this study to understand how the environment of communication (including talking about health) impact doctors' ability to find solutions and health issues to clinical problems for patients.

Participants are being asked to take part in this research study because they are either:

* A final year medical student
* OR a person willing to act out a diagnosis.

Participants will do a few tasks:

* Questionnaires: Participants will be asked to complete a questionnaire before and after a short interview. The investigators will ask participants questions to find out their general psychological traits and skills, which can affect clinical interviews. The investigators believe it should take about 10 to 15 minutes to complete the questionnaire.
* Demographic Information: The investigators will ask participants about demographics, which may include their age, gender identity, race and ethnicity.
* Interview with a medical student/patient: This will be a recorded interview between a medical student and person acting as a patient. In this meeting, they will either meet online or in person, with white noise on or off, in a brightly lit room or a regularly lit room.

  * Acting patients will be given a hypothetical condition, with a list of symptoms included. Besides this list, they will be asked to answer the medical questions as though they are themselves (e.g., height, weight)
  * Medical students will be given a list of tip questions that will help with their diagnosis.

DETAILED DESCRIPTION:
This study will link two participants: a final year medical student and an acting patient. Both will fill out consent forms outlining the study with the above purpose) standardized demographic information, and psychometric scales, including ones measuring empathy, extraversion, openness, working memory, health literacy, and fatigue. They will then be randomly put into a dyad (consisting of one medical student and one acting patient). The acting patient (who will required to be of good health- no chronic or current health issues) will be asked to pretend to have a rare or hard to diagnose health condition, having been given a document providing details of the health condition and presenting symptoms. They will be told that otherwise, they should respond to the questions as though they are themselves (for example, if the participant asked, "how tall are you", they can disclose their actual height). The medical student will be given instructions to ask all relevant questions, including a list of potential topics they should ask about, some of which are embarrassing but relevant (e.g., bowel movements).

They will then be assigned to meet the other member of their dyad in one of two conditions: online or in person (unknown to the participants). They will then act as though this is a clinical interview, to diagnose the condition. Participants will be told the investigators will be changing the lighting and background noise as a sham treatment (white noise machine and desk lamp), concealing the study's true purpose: to understand how online versus offline environments the creativity of medical providers and the tendency toward disclosure. The interview will be recorded and transcribed. At the end of the interview, participants will be debriefed by the investigators, with an explanation of the deception, and be given the ability to withdraw their data at that point.

ELIGIBILITY:
Inclusion Criteria:

* (for medical student cohort)

  1. English speaking
  2. Be enrolled in an Medical Doctorate or Doctor of Osteopathic Medicine degree
  3. Be in their final year of study
* (for the acting participant cohort)

  1. Aged 18 or older
  2. Must state they have current healthcare coverage
  3. English speaking at native fluency level

Exclusion Criteria:

* (for medical student cohort)

  1. Have previous experience as healthcare providers that is separate from their current medical training (e.g., being a nurse)
  2. Work in a technology sector
  3. Declare a conflict of interest
  4. Unable or unwilling to sign informed consent documents -(for the acting participant cohort)

  <!-- -->

  1. There is significant current or past psychiatric illness that may inhibit their ability to consent or participate (self-described)
  2. They are not willing or able to sign informed consent documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-07-29 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Creativity in medical practice (medical student- number of possible diagnoses) | From time of enrollment to end of study duration (1 hour)
  Creativity of medical practitioners will be measured using the number of possible diagnoses generated by the medical student.
Creativity in medical practice (medical student- correct diagnosis reached) | From time of enrollment to end of study duration (1 hour)
  Creativity of medical practitioners will be measured by whether or not they get the correct diagnosis.
Tendency toward disclosure by patients | From time of enrollment to end of study duration (1 hour)
  We will measure how many words the acting participants use to describe their health condition when asked an embarrassing question, without further prompting by the medical student.

CONTACTS AND LOCATIONS:
Overall Officials: Ayoub Bouguettaya, PhD, Principal Investigator — Cedars-Sinai Medical Center

IPD SHARING:
Plan to Share IPD: Yes
All data, with the exception of the interview transcripts or recordings, will be made available. This includes participant demographics with random adjustments to ensure that participant confidentiality is not compromised.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The study protocol will be public prior to the start of the study, which is anticipated to be Jul 2025
Access Criteria: This will be available on Open Science Framework as downloadable files, with the full R code for analysis and a CSV (Comma Separated Value) file of the data.
URL: https://www.osf.io/5bkwm/

REFERENCES:
- [Derived] Bouguettaya A, Aboujaoude E. The effect of remote treatment on medical provider creative thinking and patient disclosure: protocol for the MED-CREATE trial. Trials. 2025 Oct 6;26(1):389. doi: 10.1186/s13063-025-09121-0. PMID 41053846
- See also: This is the OSF link where data will be shared. The protocol is about to be submitted for peer review in an academic journal. — https://osf.io/5bkwm/